CLINICAL TRIAL: NCT00673439
Title: A Phase II Trial Using Fondaparinux in Patients With Confirmed or Suspected Heparin-Induced Thrombocytopenia (HIT)
Brief Title: Fondaparinux for the Treatment of Heparin-Induced Thrombocytopenia (HIT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated due to low accrual
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07.0100; BCC-NON-07-001 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: heparin-induced thrombocytopenia; thrombocytopenia; HIT; thrombosis; blood clot; blood thinner; anticoagulant; heparin; warfarin; fondaparinux; Arixtra
MeSH Terms: conditions — Thrombocytopenia; Thrombosis | interventions — Fondaparinux; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fondaparinux (Experimental): daily subcutaneous injection of fondaparinux (7.5-10 mg)
  Interventions: Drug: fondaparinux; Drug: warfarin

INTERVENTIONS:
Drug: fondaparinux — Dosage form: subcutaneous injection; dosage: 7.5 to 10.0 mg; frequency and duration: daily until blood test results rule out confirmed HIT - for patients with confirmed HIT, continue daily until INR (blood clotting) measurement rises to at least 2
  Other Names: Arixtra
Drug: warfarin — Dosage form: oral; dosage: 2.5 to 5.0 mg; frequency and duration: (for confirmed HIT only) once daily, to begin when blood platelet count reaches at least 100,000, and continue for approximately 4 weeks
  Other Names: Coumadin

SUMMARY:
The purpose of this study is to determine how safe and effective fondaparinux is in treating patients with suspected or confirmed heparin-induced thrombocytopenia (HIT).

DETAILED DESCRIPTION:
Currently, standard treatment of HIT involves the transition from a direct thrombin inhibitor (a type of anticoagulant or "blood thinner") to warfarin, a different type of anticoagulant. Direct thrombin inhibitors (DTIs) require IV administration and frequent blood draws for dose adjustments, which can lead to prolonged hospitalization. DTIs also affect blood test measurements, making it difficult to determine proper dosages of warfarin.

Fondaparinux is a drug that is approved by the FDA for the treatment of blood clots in deep veins and in the lungs. Fondaparinux is not FDA approved for the treatment of HIT. However, an increasing number of doctors are using fondaparinux instead of DTIs to treat HIT. Although fondaparinux appears to be more convenient and predictable than DTI medications, more research is needed to support its use as a treatment for HIT.

ELIGIBILITY:
Inclusion Criteria:

* high risk for HIT based on "Four Ts score" of 6 or more

Exclusion Criteria:

* pulmonary emboli at the time of enrollment
* arterial thrombosis at the time of enrollment
* limb threatening phlegmasia cerulea dolens at the time of enrollment
* Calculated Creatinin Clearance less than 50 ml/hr
* platelet count less than 50
* Weight less than 50 kg
* pregnancy
* allergy to fondaparinux
* bacterial endocarditis
* history of neuraxial anesthesia and post-operative indwelling epidural catheter
* active major bleeding (hemodynamically significant or requiring transfusions)
* inability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, MSPH, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fondaparinux
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fondaparinux
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  Over 18 years of age | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Clinically Significant Bleeding
Description: Clinically significant bleed is defined as Hemodynamically Significant Bleeding or Requiring Blood Transfusions While Being Treated With Fondaparinux
Time Frame: 4 weeks after INR reaches 2 or more
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: the Incidence of Venous or Thrombotic Events After Starting Treatment With Fondaparinux
Time Frame: 4 weeks after INR reaches 2 or more
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Arm/Group | Daily Subcutaneous Injection of Fondaparinux (7.5-10 mg)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Study terminated, results data not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No